CLINICAL TRIAL: NCT01265550
Title: CSP #573 - A Randomized Trial of Medical and Surgical Treatments for Patients With GERD Symptoms That Are Refractory to Proton Pump Inhibitors
Brief Title: A Randomized Trial of Medical and Surgical Treatments for Patients With GERD Symptoms That Are Refractory to Proton Pump Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 573
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Fundoplication; Baclofen; Desipramine

STUDY DESIGN:
Masking Description: Partial Double Blind (Medical Treatment Groups)
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Medical Treatment Group (Other): Omeprazole or Omeprazole + baclofen or Omeprazole + desipramine
  Interventions: Drug: baclofen; Drug: Desipramine
- Surgical Treatment Group (Other): Laparoscopic nissen fundoplications
  Interventions: Device: Nissen fundoplication
- Placebo Medical Treatment Group (Other): Omeprazole + placebo
  Interventions: Drug: baclofen; Drug: Desipramine

INTERVENTIONS:
Device: Nissen fundoplication — laparoscopic antireflux surgery
  Arms: Surgical Treatment Group
Drug: baclofen — Baclofen will be prescribed in a dose of 5 mg three times a day (TID) with meals.
  The dose of baclofen will be increased by 5 mg TID every week until a total dose of 20 mg TID has been achieved.
  Arms: Medical Treatment Group; Placebo Medical Treatment Group
Drug: Desipramine — Dose of 25 mg at bedtime (HS) for 1 week, then 50 mg HS for 1 week, then 100 mg HS until the next quarterly visit.
  Arms: Medical Treatment Group; Placebo Medical Treatment Group

SUMMARY:
Background: Gastroesophageal reflux disease (GERD), which affects at least 20% of adult Americans, may be especially common and severe in Veteran patients. Proton pump inhibitors (PPIs), which block gastric acid production, are the most effective medications for GERD, and the VA spends more than $177 million each year on outpatient PPI prescriptions. PPIs do not prevent the reflux of non-acidic material and do not completely eliminate esophageal acid exposure, however, and bothersome GERD symptoms persist in approximately 40% of patients treated with PPIs. Recent studies using the new technique of esophageal pH/ impedance monitoring, which detects the reflux of both acidic and non-acidic materials, have shown that PPI-resistant GERD symptoms correlate with episodes of reflux (acidic and/or non-acidic) in approximately one-half of patients. For those patients, an antireflux operation might relieve symptoms and obviate the expense of ineffective PPI therapy, but the efficacy of modern, laparoscopic fundoplication in this regard is not clear. For patients with PPI-resistant GERD symptoms, furthermore, the efficacy of medications that that can prevent gastroesophageal reflux (e.g. baclofen) or diminish pain of esophageal origin (e.g. neurotropic agents like desipramine) also is not clear. Study Hypothesis: Laparoscopic antireflux surgery (Nissen fundoplication) is superior to medical therapy (PPIs plus baclofen and desipramine) for GERD patients who, while on PPIs, have persistent episodes of heartburn that are associated with reflux episodes or with abnormal esophageal acid exposure by esophageal pH/impedance monitoring.

Study Goals: The primary goal is to compare the efficacy of laparoscopic Nissen fundoplication and medical therapy (PPIs plus baclofen and desipramine) for GERD patients who, while on PPIs, have persistent episodes of heartburn that are associated with reflux episodes or with abnormal esophageal acid exposure by esophageal pH/impedance monitoring, and to compare the efficacy of each therapy with placebo. Secondary goals are: 1) To determine the frequency with which non-GERD disorders underlie "PPI failure," 2) To determine the frequency of functional gastrointestinal symptoms, anxiety and depression in patients who have persistent heartburn while on PPIs, 3) To determine whether functional gastrointestinal symptoms, anxiety and depression is associated with the outcomes of medical and surgical therapies, and 4) To determine whether the outcome of Nissen fundoplication is associated with adherence to technical aspects of the operation.

Study Design: Up to 16 VA medical centers, there will be a 30-month recruitment period to enroll 108 patients with heartburn that is refractory to PPI therapy. Patients will have their baseline GERD symptoms scored using the GERD Health-Related Quality of Life (GERD-HRQL) index, and will have endoscopy, esophageal manometry and esophageal pH/impedance monitoring while on PPI therapy. Patients who have episodes of heartburn that are associated with reflux episodes or with abnormal esophageal acid exposure by esophageal pH/impedance monitoring will be randomized to one of three treatment groups: Surgical Treatment (laparoscopic Nissen fundoplication), Active Medical Treatment (omeprazole and baclofen initially; desipramine for baclofen failures) or Placebo Medical Treatment (omeprazole, placebo baclofen, placebo desipramine). All patients will have quarterly clinic visits for symptom scoring and laboratory testing. At one year, patients will have a final symptom scoring and repeat endoscopy, esophageal manometry and esophageal pH/impedance monitoring. Treatment success will be defined as 50% improvement in the GERD-HRQL score at 12 months. Patients also will complete the Hospital Anxiety and Depression Scale (HADS), Rome III Functional GI Disorders Questionnaire and the Short-Form Health Survey (SF-36) at baseline and one year. The results will be correlated with treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* History of heartburn (defined as a burning sensation in the retrosternal area of the chest) that is refractory to antisecretory medications
* Initial GERD-HRQL:

  * Total score must be at least 6 and at least one of the six heartburn questions must be scored at least 2
* GERD-HRQL after two weeks of treatment with omeprazole:

  * Total score must be >50% of the initial GERD-HRQL score and at least one of the six heartburn questions must be scored at least 2
* Either or both of the following by baseline esophageal pH/multichannel intraluminal impedance (MII) monitoring in patients on omeprazole 20 mg two times a day (BID):

  * Positive symptom association probability (SAP) (>95%) for acid reflux, non-acid reflux or all reflux.
  * Abnormal acid reflux (esophageal pH<4 for at least 4.2% of the 24-hour monitoring period)

Exclusion Criteria:

* Patients who do not have heartburn, defined as a burning sensation in the chest
* Patients unwilling or unable to provide informed consent
* Pregnancy or women unwilling to use effective contraception
* Age <18 or >70 years
* History of surgery on the stomach or esophagus
* History of seizure disorder
* History of heart block
* Allergy to or previous inability to tolerate study medications (omeprazole, baclofen, desipramine)
* Esophageal varices
* Cirrhosis
* Co-morbidity of sufficient severity to preclude elective surgery (e.g. pulmonary, cardiac, renal, liver disease)
* History of disorders that can cause medically-refractory "GERD symptoms" (eosinophilic esophagitis, neoplasms of the upper gastrointestinal tract, gastroparesis, achalasia)
* Myocardial infarction within the past 6 months
* History of schizophrenia
* Current use of clopidogrel
* Patients who have a contraindication to omeprazole or baclofen or who require therapy with a medication that has a clinically important drug interaction with omeprazole or baclofen.
* Patients who, in the judgment of the PI, are not suitable candidates for therapy with a study medication (omeprazole, baclofen, desipramine)
* Initial GERD-HRQL score: Total score <6 and/or all heartburn scores <2
* Inability to tolerate omeprazole during the 2-week treatment phase (before randomization)
* GERD-HRQL after two weeks of treatment with omeprazole: Total score less than or equal to 50% of initial GERD-HRQL score and/or all heartburn scores <2
* Laboratory abnormalities including:

  * Platelet count <100,000
  * international normalized ratio (INR) >1.5 (off anticoagulants)
  * Serum creatinine >2.0 mg per deciliter
* Endoscopic abnormalities including:

  * Los Angeles Classification of Oesophagitis (LA grade) C or D reflux esophagitis
  * Active ulceration of the esophagus that is not due to reflux esophagitis
  * Candida esophagitis
  * Esophageal varices
  * Active ulceration of the stomach and/or duodenum
  * Neoplasm of the esophagus, stomach or duodenum
  * Gastric outlet obstruction
  * Eosinophilic esophagitis at least (15 eosinophils per high power field in any esophageal biopsy specimen)
* Manometric abnormalities including:

  * Achalasia
  * Complete aperistalsis
* Negative SAP ( 95%) for acid reflux, non-acid reflux and all reflux on baseline combined esophageal pH/MII monitoring and normal acid reflux (esophageal pH<4 for <4.2% of the 24-hour monitoring period)
* Study surgeon identifies a contraindication to laparoscopic Nissen fundoplication
* Morbid obesity (BMI at least 40)
* Large paraesophageal hernia

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 366 (Actual)
Dates: Start 2012-08-13 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Spechler, MD, Study Chair — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (15):
- United States (15):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spechler SJ, Hunter JG, Jones KM, Lee R, Smith BR, Mashimo H, Sanchez VM, Dunbar KB, Pham TH, Murthy UK, Kim T, Jackson CS, Wallen JM, von Rosenvinge EC, Pearl JP, Laine L, Kim AW, Kaz AM, Tatum RP, Gellad ZF, Lagoo-Deenadayalan S, Rubenstein JH, Ghaferi AA, Lo WK, Fernando RS, Chan BS, Paski SC, Provenzale D, Castell DO, Lieberman D, Souza RF, Chey WD, Warren SR, Davis-Karim A, Melton SD, Genta RM, Serpi T, Biswas K, Huang GD. Randomized Trial of Medical versus Surgical Treatment for Refractory Heartburn. N Engl J Med. 2019 Oct 17;381(16):1513-1523. doi: 10.1056/NEJMoa1811424. PMID 31618539

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Treatment Group; Placebo Medical Treatment Group: baclofen: Baclofen will be prescribed in a dose of 5 mg three times a day (TID) with meals.
  The dose of baclofen will be increased by 5 mg TID every week until a total dose of 20 mg TID has been achieved.
  Desipramine: Dose of 25 mg at bedtime (HS) for 1 week, then 50 mg HS for 1 week, then 100 mg HS until the next quarterly visit.
- All Enrolled: All patients consented.
Period: Pre Randomization
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group | All Enrolled
Started | 0 | 0 | 0 | 366
Completed | 0 | 0 | 0 | 78
Not Completed | 0 | 0 | 0 | 288
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 70
Not completed — Technical Exclusions | 0 | 0 | 0 | 54
Not completed — GERD, PPI-Responsive | 0 | 0 | 0 | 42
Not completed — Non-GERD organic disorders | 0 | 0 | 0 | 23
Not completed — Functional heartburn | 0 | 0 | 0 | 99
Period: Post Randomization
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group | All Enrolled
Started | 25 | 27 | 26 | 0
Completed | 10 | 19 | 6 | 0
Not Completed | 15 | 8 | 20 | 0

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized: Subset of all enrolled participants who did not end up being randomized to the study.
- Total: Total of all reporting groups
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group | Not Randomized | Total
Number analyzed (Participants) | 25 | 27 | 26 | 288 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing data
  years
    number analyzed (Participants) | 25 | 27 | 26 | 280 | 358
    (all) | 43.9 (12.2) | 44.9 (11.8) | 47.2 (11.7) | 49.3 (12.2) | 45.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data.
  Participants
    number analyzed (Participants) | 25 | 27 | 26 | 279 | 357
    Female | 7 | 4 | 3 | 63 | 77
    Male | 18 | 23 | 23 | 216 | 280
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Missing data.
  Participants
    number analyzed (Participants) | 25 | 27 | 26 | 279 | 357
    Hispanic or Latino | 4 | 7 | 2 | 40 | 53
    Not Hispanic or Latino | 21 | 20 | 23 | 230 | 294
    Unknown or Not Reported | 0 | 0 | 1 | 9 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 25 | 27 | 26 | 279 | 357
    American Indian or Alaska Native | 0 | 0 | 0 | 3 | 3
    Asian | 0 | 0 | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
    Black or African American | 2 | 2 | 5 | 54 | 63
    White | 20 | 17 | 17 | 183 | 237
    More than one race | 2 | 2 | 2 | 16 | 22
    Unknown or Not Reported | 1 | 6 | 1 | 21 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving at Least a 50% Improvement in the Gastroesophageal Reflux Disease Health-related Quality of Life Index (GERD-HRQL) From Baseline to 12 Months
Description: Success; ≥50% improvement in the baseline GERD-HRQL score at 12 months.
  Failure; <50% improvement in the baseline GERD-HRQL score at 12 months or:
  1. For patients randomized to Surgical Treatment: a.<50% improvement in the baseline GERD-HRQL score and/or persistent heartburn of sufficient severity to warrant treatment with any antisecretory medication, antireflux medication or neurotropic medication at any quarterly clinic visit.
  2. For patients randomized to Active Medical or Placebo Medical Treatment:
     a.inability to tolerate both study medications or b.For patients treated with desipramine, i.<50% improvement in baseline GERD-HRQL score symptom after at least 10 weeks of treatment with the second drug at any quarterly clinic visit. c.For patients in whom desipramine is contraindicated,i.<50% improvement in baseline GERD-HRQL score symptom after at least 10 weeks of treatment with baclofen or its corresponding placebo at any quarterly clinic visit.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 25 | 27 | 26
Participants | 7 | 18 | 3

2. Secondary Outcome: Number of Enrolled Participants With Esophageal Ulceration.
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for esophageal ulceration.
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 216
Participants | 0

3. Secondary Outcome: Number of Enrolled Participants With Reflux Esophagus.
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for reflux esophagus.
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 216
Participants | 4

4. Secondary Outcome: Number of Enrolled Participants With Eosinophilic Esophagitis
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for eosinophilic esophagitis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 215
Participants | 16

5. Secondary Outcome: Number of Enrolled Participants With Active Ulceration of the Stomach and/or Duodenum.
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for active ulcerations of the stomach and/or duodenum
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 216
Participants | 3

6. Secondary Outcome: Number of Enrolled Participants With Neoplasm of the Esophagus, Stomach or Duodenum
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for neoplasm of the esophagus, stomach or duodenum
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 216
Participants | 0

7. Secondary Outcome: Number of Enrolled Participants With Candida Esophagitis.
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for candida esophagitis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 216
Participants | 3

8. Secondary Outcome: Number of Enrolled Participants With Gastric Outlet Obstruction
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for gastric outlet obstruction
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 216
Participants | 0

9. Secondary Outcome: Number of Enrolled Participants With Achalasia
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for achalasia
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 212
Participants | 2

10. Secondary Outcome: Number of Enrolled Participants With Aperistalsis
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for aperistalsis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 212
Participants | 0

11. Secondary Outcome: Number of Enrolled Participants With Distal Esophageal Spasm
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for distal esophageal spasm
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 212
Participants | 3

12. Secondary Outcome: Number of Enrolled Participants With Nutcracker Esophagus
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for nutcracker esophagus
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 32
Participants | 2

13. Secondary Outcome: Number of Enrolled Participants With Ineffective Esophageal Motility
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for ineffective esophageal motility
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 33
Participants | 1

14. Secondary Outcome: Number of Enrolled Participants With Rapid Contraction
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for rapid contraction
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 93
Participants | 2

15. Secondary Outcome: Number of Enrolled Participants With Hypertensive Peristalsis
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for hypertensive peristalsis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 93
Participants | 3

16. Secondary Outcome: Number of Enrolled Participants With Jackhammer Esophagus
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for jackhammer esophagus
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 93
Participants | 8

17. Secondary Outcome: Number of Enrolled Participants With Weak Peristalsis I
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for weak peristalsis I
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 93
Participants | 10

18. Secondary Outcome: Number of Enrolled Participants With Weak Peristalsis II
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for weak peristalsis II
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 93
Participants | 9

19. Secondary Outcome: Number of Enrolled Participants With Anxiety and/or Depression
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for anxiety and/or depression
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 272
Participants | 125

20. Secondary Outcome: Number of Enrolled Participants With Functional Heartburn
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for functional heartburn
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 274
Participants | 221

21. Secondary Outcome: Number of Enrolled Participants With Functional Chest Pain of Presumed Esophageal Origin
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for functional chest pain of presumed esophageal origin
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 276
Participants | 13

22. Secondary Outcome: Number of Enrolled Participants With Functional Dysphagia
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for functional dysphagia
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 277
Participants | 7

23. Secondary Outcome: Number of Enrolled Participants With Globus
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for globus
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 278
Participants | 0

24. Secondary Outcome: Number of Enrolled Participants With Belching Disorders
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for belching disorders
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 273
Participants | 130

25. Secondary Outcome: Number of Enrolled Participants With Chronic Idiopathic Nausea
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for chronic idiopathic nausea
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 273
Participants | 51

26. Secondary Outcome: Number of Enrolled Participants With Functional Vomiting
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for functional vomiting
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 276
Participants | 32

27. Secondary Outcome: Number of Enrolled Participants With Cyclic Vomiting Syndrome
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for cyclic vomiting syndrome
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 276
Participants | 86

28. Secondary Outcome: Number of Enrolled Participants With Irritable Bowel Syndrome
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for irritable bowel syndrome
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 277
Participants | 152

29. Secondary Outcome: Number of Enrolled Participants With Functional Bloating
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for functional bloating
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 277
Participants | 8

30. Secondary Outcome: Number of Enrolled Participants With Functional Diarrhea
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for functional diarrhea
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 271
Participants | 4

31. Secondary Outcome: Number of Enrolled Participants With Unspecified Functional Bowel Disorder
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for unspecified functional bowel disorder
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 278
Participants | 56

32. Secondary Outcome: Number of Enrolled Participants With Functional Gallbladder Disorder
Time Frame: Screening
Population: The Overall number of participants analyzed represents those Enrolled Participants who were evaluated for functional gallbladder disorder
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 278
Participants | 1

33. Secondary Outcome: Number of Successful Participants With Anxiety and/or Depression.
Description: Association between anxiety and/or depression (GAD-7 and PHQ-9) and the outcome of medical and surgical treatments (success or failure) will be evaluated.
Time Frame: 12 months
Population: Number of treatment successes.
Measure: Count of Participants; unit: Participants
Groups:
- Medical Treatment Group: Omeprazole + baclofen or Omeprazole + desipramine
  baclofen: Baclofen will be prescribed in a dose of 5 mg three times a day (TID) with meals.
  The dose of baclofen will be increased by 5 mg TID every week until a total dose of 20 mg TID has been achieved.
  Desipramine: Dose of 25 mg at bedtime (HS) for 1 week, then 50 mg HS for 1 week, then 100 mg HS until the next quarterly visit.
- Placebo Medical Treatment Group: Omeprazole + placebo
  baclofen: Baclofen will be prescribed in a dose of 5 mg three times a day (TID) with meals.
  The dose of baclofen will be increased by 5 mg TID every week until a total dose of 20 mg TID has been achieved.
  Desipramine: Dose of 25 mg at bedtime (HS) for 1 week, then 50 mg HS for 1 week, then 100 mg HS until the next quarterly visit.
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 2 | 5 | 0

34. Secondary Outcome: Number of Successful Participants With Functional Heartburn
Description: Presence of functional heartburn as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 7 | 14 | 3

35. Secondary Outcome: Number of Successful Participants With Functional Chest Pain of Presumed Esophageal Origin
Description: Presence of functional chest pain of presumed esophageal origin as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 0 | 0 | 0

36. Secondary Outcome: Number of Successful Participants With Functional Dysphagia
Description: Presence of functional dysphagia as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 0 | 0 | 0

37. Secondary Outcome: Number of Successful Participants With Globus
Description: Presence of globus as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 0 | 0 | 0

38. Secondary Outcome: Number of Successful Participants With Belching Disorders
Description: Presence of belching disorders as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 3 | 12 | 2

39. Secondary Outcome: Number of Successful Participants With Chronic Idiopathic Nausea
Description: Presence of chronic idiopathic nausea as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 0 | 3 | 0

40. Secondary Outcome: Number of Successful Participants With Functional Vomiting
Description: Presence of functional vomiting as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 1 | 1 | 1

41. Secondary Outcome: Number of Successful Participants With Cyclic Vomiting Syndrome
Description: Presence of cyclic vomiting syndrome as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 1 | 7 | 1

42. Secondary Outcome: Number of Successful Participants With Irritable Bowel Syndrome
Description: Presence of irritable bowel syndrome as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 3 | 10 | 3

43. Secondary Outcome: Number of Successful Participants With Functional Bloating
Description: Presence of functional bloating as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 1 | 1 | 0

44. Secondary Outcome: Number of Successful Participants With Functional Diarrhea
Description: Presence of functional diarrhea as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 0 | 0 | 0

45. Secondary Outcome: Number of Successful Participants With Unspecified Functional Bowel Disorder
Description: Presence of unspecified functional bowel disorder as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes.
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 2 | 5 | 0

46. Secondary Outcome: Number of Successful Participants With Functional Gallbladder Disorder
Description: Presence of functional gallbladder disorder as assessed by the ROME III functional GI disorders questionnaire.
Time Frame: 12 months
Population: Number of treatment successes
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group
Number analyzed (Participants) | 7 | 18 | 3
Participants | 0 | 0 | 0

47. Secondary Outcome: Number of Successful Surgery Participants With Dissection of Distal Esophagus to Obtain at Least 2.5cm of Tension-free, Intra-abdominal Esophagus Performed.
Time Frame: 12 months
Population: Surgical participants with at least 50% improvement in the baseline GERD-HRQL score at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Treatment Group
Number analyzed (Participants) | 18
Participants | 18

48. Secondary Outcome: Number of Successful Surgery Participants With Complete Mobilization of the Fundus, to Include All Short Gastric and Posterior Gastric Vessels to the Base of the Left Crus Performed.
Time Frame: 12 months
Population: Surgical participants with at least 50% improvement in the baseline GERD-HRQL score at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Treatment Group
Number analyzed (Participants) | 18
Participants | 18

49. Secondary Outcome: Number of Successful Surgery Participants With Closure of the Crura With Non-absorbable Suture to be Snug With a Dilator of at Least 56 French Diameter Performed.
Time Frame: 12 months
Population: Surgical participants with at least 50% improvement in the baseline GERD-HRQL score at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Treatment Group
Number analyzed (Participants) | 18
Participants | 14

50. Secondary Outcome: Number of Successful Surgery Participants With Passage of an Esophageal Dilator of at Least 56 French Diameter Performed.
Time Frame: 12 months
Population: Surgical participants with at least 50% improvement in the baseline GERD-HRQL score at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Treatment Group
Number analyzed (Participants) | 18
Participants | 14

51. Secondary Outcome: Number of Successful Surgery Participants With Fundoplication Between 1.5 and 2.5cm in Length Performed.
Time Frame: 12 months
Population: Surgical participants with at least 50% improvement in the baseline GERD-HRQL score at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Treatment Group
Number analyzed (Participants) | 18
Participants | 18

52. Secondary Outcome: Number of Successful Surgery Participants With Fundoplication Placed Above the Epiphrenic Fat Pad, Using 3 Sutures Performed.
Time Frame: 12 months
Population: Surgical participants with at least 50% improvement in the baseline GERD-HRQL score at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Treatment Group
Number analyzed (Participants) | 18
Participants | 18

53. Secondary Outcome: Number of Successful Surgery Participants With Fundoplication Secured to Esophagus With at Least Two Sutures Performed.
Time Frame: 12 months
Population: Surgical participants with at least 50% improvement in the baseline GERD-HRQL score at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Treatment Group
Number analyzed (Participants) | 18
Participants | 18

54. Secondary Outcome: Number of Successful Surgery Participants With Fundoplication Floppiness Demonstrated by Passing a Grasper Between Fundoplication and Dilator-filled Esophagus Performed.
Time Frame: 12 months
Population: Surgical participants with at least 50% improvement in the baseline GERD-HRQL score at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Treatment Group
Number analyzed (Participants) | 18
Participants | 15

ADVERSE EVENTS:
Time Frame: From consent to subject termination, up to 14 months.
Description: Events reported in the all enrolled column were events that occurred prior to randomization. Events that occurred after randomization are reported under the respective treatment group.
Arm/Group | Medical Treatment Group | Surgical Treatment Group | Placebo Medical Treatment Group | All Enrolled
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27 | 0/26 | 0/288
Serious Adverse Events (participants affected / at risk) | 4/25 | 4/27 | 3/26 | 15/366
Other Adverse Events (participants affected / at risk) | 18/25 | 17/27 | 18/26 | 79/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Treatment Group (N=25) | Surgical Treatment Group (N=27) | Placebo Medical Treatment Group (N=26) | All Enrolled (N=366)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture of penis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Violence-related symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporal arteritis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Treatment Group (N=25) | Surgical Treatment Group (N=27) | Placebo Medical Treatment Group (N=26) | All Enrolled (N=366)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 8 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 4 (5) | 1 (1) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (6)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (2) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laboratory test (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood HIV RNA increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dacryoadenitis acquired (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes